CLINICAL TRIAL: NCT01722708
Title: Comparison Between Oral Clindamycin Vs Metronidazole for the Treatment of Abnormal Vaginal Flora in High Risk Pregnancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0012-12-EMC
Record Dates: First submitted 2012-10-28; First posted 2012-11-07 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Abnormal Vaginal Flora; Clindamycin Vs Metronidazole; High Risk Pregnancies for Preterm Labor
Keywords: Abnormal vaginal flora; clindamycin Vs metronidazole; High risk pregnancies for preterm labor; Preterm labor; Late abortion; bacterial vaginosis
MeSH Terms: conditions — Obstetric Labor, Premature; Vaginosis, Bacterial | interventions — Clindamycin; Metronidazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- clindamycin (Experimental)
  Interventions: Drug: Clindamycin
- metronidazole (Experimental)
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Clindamycin — Oral clindamycin 300 Milligrams*2/Day for a week
  Arms: clindamycin
Drug: Metronidazole — Oral metronidazole 500 Milligrams*2/Day for a week
  Arms: metronidazole

SUMMARY:
Abnormal vaginal flora is a risk factor for preterm labor. Therefore, in high risk pregnancies for preterm labor the diagnosis and treatment of abnormal flora is indicated. Clindamycin and metronidazole given orally are both acceptable treatments in these cases. The purpose of this study is to compare the effectiveness of Clindamycin Vs metronidazole for the treatment of abnormal vaginal flora in high risk pregnancies. For this purpose, pregnant women who are considered high risk for preterm labor and were diagnosed with abnormal vaginal flora will be randomly treated either with clindamycin or metronidazole. Eradication of the abnormal flora and adverse effects will be monitored and compared

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at increased risk for preterm labor (preterm cervical effacement, preterm uterine contractions, twins pregnancy, vaginal bleeding, past preterm delivery)
* Age above 18 years

Exclusion Criteria:

* Known allergy to the tested antibiotics
* Antibacterial treatment in the week before the vaginal culture was taken
* preterm premature rupture of membranes

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy between oral Clindamycin Vs Metronidazole in the eradication of abnormal vaginal flora | Primary outcome will be assessed by taking a vaginal culture sample a week after one-week antibacterial treatment

SECONDARY OUTCOMES:
The prevalence of adverse effects | During the antibacterial treatment which is 1 week of therapy
The prevalence of late abortions and preterm deliveries | From date of randomization until the date of delivery or abortion, assessed up to 28 weeks
Assessing the correlation between Nugent score , physical examination and Ph indicators | The outcome is assessed after the diagnosis of abnormal vaginal flora is made at 14-26 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Zohar Nachum, MD, Principal Investigator — Departement of obstetric and gynecology, HaEmek medical center, Afula, Israel
Locations (2):
- Israel (2):
  - Departement of obstetric and gynecology, Poriya Medical Center, Tiberias, Israel
  - Departement of obstetric and gynecology, HaEmek medical center, Afula